CLINICAL TRIAL: NCT05025787
Title: EN20-01: A 24 Week Study to Evaluate the Safety and Efficacy of CNTX-6970 in Subjects With Moderate to Severe Knee Osteoarthritis Pain.
Brief Title: A Study to Evaluate the Safety and Efficacy of CNTX-6970 in Subjects With Knee Osteoarthritis Pain.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maurizio Fava, MD (Other)
Responsible Party: Sponsor-Investigator, Maurizio Fava, MD, Psychiatrist in Chief, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021p002273 (EN20-01)
Record Dates: First submitted 2021-08-16; First posted 2021-08-27 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The study will employ a randomized, allocation-concealed, multicenter, placebo-controlled, multi-period crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding of the randomization assignment from trial subjects, staff from the Clinical Sites, CCC, and DCC will be ensured through the use of the IXRS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 300mg BID CNTX-6970, Then Placebo (Experimental): Participants initially received 300 mg BID of CNTX-6970 for 6 weeks (Block 1, Period 1). Following this, they were administered matching placebo BID for another 6 weeks (Block 1, Period 2). After a total of 12 weeks, participants received 300 mg BID of CNTX-6970 again for 6 weeks (Block 2, Period 1). Finally, after 18 weeks of total treatment, participants received a matching placebo for an additional 6 weeks (Block 2, Period 2), completing a 24-week study period.
  Interventions: Drug: CNTX-6970; Drug: Placebo
- Placebo, then 300 mg BID CNTX-6970 (Placebo Comparator): Participants initially received placebo BID for 6 weeks (Block 1, Period 1). Following this, they were administered 300 mg CNTX-9670 BID for another 6 weeks (Block 1, Period 2). After a total of 12 weeks, participants received placebo BID again for 6 weeks (Block 2, Period 1). Finally, after 18 weeks of total treatment, participants received a 300 mg CNTX-6970 BID for an additional 6 weeks (Block 2, Period 2), completing a 24-week study period.
  Interventions: Drug: CNTX-6970; Drug: Placebo

INTERVENTIONS:
Drug: CNTX-6970 — CNTX-6970, a novel potent antagonist of CCR2 with lesser effects on CCR5, is being developed as a new treatment for chronic pain, including painful osteoarthritis of the knee.
Drug: Placebo — BID
  Other Names: Matching Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of CNTX-6970 for the treatment of pain related to OA of the knee compared to placebo. CNTX-6970 is being developed as a new treatment for chronic pain, including painful osteoarthritis of the knee.

DETAILED DESCRIPTION:
The study will employ a randomized, allocation-concealed, multicenter, placebo-controlled, multi-period crossover design (Schmid et al, 2018). This multi-period crossover randomized, controlled trial allows comparability and assessment of efficacy through repeated exposures within each subject to the active treatment and a control (placebo) in randomized sequence. Such multi-period crossover designs are ideal for treatments with rapid onset of action and short half-life such as the asset under study here. We have strived to minimize the complexity of this powerful design by using only 2 blocks with 2 periods each. The modest additional complexity of the proposed multi-period crossover design, compared to a parallel-groups design, is justified by the marked improvement in efficiency. The gains in efficiency afforded by the multi-period crossover design allow a substantial reduction in sample size without sacrificing statistical power.

The trial will compare an active treatment vs. placebo. Each block will consist of two treatment periods with each period lasting 6 weeks. Treatment assignments (active drug versus placebo) will be randomized for each patient to the two periods within each block. The period length of 6 weeks was chosen based on several considerations: (i) Most efficacious analgesic drugs demonstrate separation from placebo by 6 weeks; (ii) The decision to move CNTX-6970 forward to Phase 3 will require a clinically meaningful separation from placebo by 6 weeks; (iii) In this Phase 2 study, implementing a treatment block longer than 6 weeks would make the overall design more challenging and burdensome by extending the duration of overall testing beyond 6 months; (iv).

In this study, the placebo will consist of inactive tablets identical to the active treatment tablets. Treatment assignments (active drug versus placebo) will be randomized for each patient to the two treatment periods within each block.

ELIGIBILITY:
A subject will be eligible for study participation if they meet all of the following criteria:

1. Individuals between 40 and 90 years of age (inclusive) at the time of the Screening Visit.
2. Willing to use a mobile smart device during the study period. Individuals who do not have access to a mobile device will be provided with one for the duration of the study and trained in its use.
3. Can understand the nature of the study and protocol requirements and is willing to comply with study drug administration requirements and discontinue prohibited concomitant medications.
4. Radiography of both knees with a posterior-anterior, fixed-flexion view taken during the Screening visit. The Index knee must show evidence of chronic OA with a K-L Grading Scale of 1, 2, 3, or 4. Such evidence will be provided by a central reading of the radiography of both knees from an expert radiologist of the CCC of EPPIC-Net.
5. Moderate to severe pain in the Index knee associated with OA and stable for a minimum of 6 months prior to Screening in the opinion of the investigator.
6. Confirmation of OA of the index knee: American College of Rheumatology (ACR) diagnostic criteria.
7. Subjects must have failed 2 or more prior therapies. Failure is deemed to be inadequate relief in the opinion of the investigator.
8. Body mass index (BMI) of ≤ 40 kg/m2.
9. Willing to refrain from illicit drug use during the study, and to have illicit drug testing at screening and at later time points.

A subject will be excluded from the study if they meet any of the following criteria:

1. Any form of joint replacement surgery, open surgery, or arthroscopic surgery of the index knee/knee joint with 12 months of Screening.
2. Any painful condition(s) of the index knee due to disease other than OA. For example, periarticular or referred pain involving the index knee, or from joint disease other than OA associated with the index knee.
3. Other chronic pain anywhere in the lower extremities (e.g. hips, legs, feet) that is equal or greater in intensity or impairment than index knee pain or that requires the use of analgesic medications. This includes radicular low back pain with radiation to the knee.
4. Documented history of neuropathic arthropathy in the knee.
5. Significant instability (e.g., cruciate ligament tear or rupture or previous repair) within the past 5 years or current misalignment (>10 degrees varus or valgus) of the index knee.
6. Plans to have surgery, invasive procedures, or intra-articular (IA) injections of the index knee or procedure or surgery otherwise contraindicated for study participation while in the study.

   a. Concomitant Medications for Pain - i. Continuous use of one of the following medications prescribed for pain: tramadol, gabapentin, duloxetine, pregabalin, milnacipran, or tricyclic antidepressants that is:
   1. chronic for at least 12 weeks; and
   2. at a stable dose for at least 4 weeks before Screening ii. Intermittent use of opioids that is:

   <!-- -->

   1. ongoing for at least 4 weeks before Screening;
   2. at a frequency no more than 4 days/week; and
   3. not be taken within 24 hours of a study visit

   iii. As needed use of acetaminophen iv. Continuous use of medical marijuana (or equivalent) that is chronic for at least 12 weeks and at a stable dose for 4 weeks v. Topical creams (includes CBD topicals)
   1. Continuous use allowed if chronic and stable for at least 12 weeks
   2. Intermittent use allowed if at a frequency of no more than 4 days/week

   b. Concomitant Medications for Non-Pain Indications That May Impact Pain - i. Continuous use of medication for non-pain indications that are known to potentially impact pain, e.g. duloxetine for depression, that is at a stable dose for at least 12 weeks prior to Screening.

   ii. Low-dose aspirin for the purposes of heart disease prophylaxis
7. Corticosteroid injection in the index knee within 30 days of Screening or during study participation (unless the injectable is a long-acting agent such as triamcinolone acetonide extended-release injectable suspension (Zilretta) in which case the injection cannot be within 90 days of screening).
8. Received IA viscosupplementation (e.g., Synvisc®, Hyalgan®) within 90 days of Screening.

10. Use of an investigational medication within 30 days of Screening, or 5 pharmacokinetic or pharmacodynamic half-lives (whichever is longer) or scheduled to receive such an agent while participating in the current study.

11. Current therapy with any immunosuppressive therapy, including corticosteroids (>5 mg/day of prednisone).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hosptial
Locations (16):
- United States (16):
  - University of California San Diego, La Jolla, California
  - University of California- Davis, Sacramento, California
  - University of Florida, Gainesville, Florida
  - M&M Clinical Trials, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Healthcare Research Network, Hazelwood, Missouri
  - New York University Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Center for Clinical Research, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UTsouthwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington
  - University of Wisconsin- Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The EPPIC-Net DCC's NYU Center for Biospecimen Research and Development (CBRD) will store and manage biological samples (biosamples) collected in this clinical trial. The samples will be used for the present study and also for potential future research as permitted by the study-specific informed consent form. Biosamples stored for this study may include, but are not limited to: whole blood, plasma, stool, synovial fluid, and/or derivatives of these specimens. The samples will be stored only for the period defined in the informed consent form, which may be indefinite. Biospecimens may be shared in accordance with the protocol-defined data and sample sharing plan and the informed consent form.
  Biosamples will be documented in LabVantage, a secure network linking biospecimens to corresponding clinical and pathological data. LabVantage does not include any identifying personal health information (PHI). The CBRD and LabVantage meet all General Lab Protocol (GLP) and FDA guidelines.
Supporting Information: ICF

REFERENCES:
- [Background] Arnold SE, Betensky RA. Multicrossover Randomized Controlled Trial Designs in Alzheimer Disease. Ann Neurol. 2018 Aug;84(2):168-175. doi: 10.1002/ana.25280. Epub 2018 Aug 29. PMID 30014506
- [Background] Arroll B, Goodyear-Smith F, Crengle S, Gunn J, Kerse N, Fishman T, Falloon K, Hatcher S. Validation of PHQ-2 and PHQ-9 to screen for major depression in the primary care population. Ann Fam Med. 2010 Jul-Aug;8(4):348-53. doi: 10.1370/afm.1139. PMID 20644190
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Bhangoo S, Ren D, Miller RJ, Henry KJ, Lineswala J, Hamdouchi C, Li B, Monahan PE, Chan DM, Ripsch MS, White FA. Delayed functional expression of neuronal chemokine receptors following focal nerve demyelination in the rat: a mechanism for the development of chronic sensitization of peripheral nociceptors. Mol Pain. 2007 Dec 12;3:38. doi: 10.1186/1744-8069-3-38. PMID 18076762
- [Background] Boakye M, Harkema S, Ellaway PH, Skelly AC. Quantitative testing in spinal cord injury: overview of reliability and predictive validity. J Neurosurg Spine. 2012 Sep;17(1 Suppl):141-50. doi: 10.3171/2012.5.AOSPINE1296. PMID 22985380
- [Background] Bruehl S, Liu X, Burns JW, Chont M, Jamison RN. Associations between daily chronic pain intensity, daily anger expression, and trait anger expressiveness: an ecological momentary assessment study. Pain. 2012 Dec;153(12):2352-2358. doi: 10.1016/j.pain.2012.08.001. Epub 2012 Aug 30. PMID 22940462
- [Background] Buckner JD, Crosby RD, Silgado J, Wonderlich SA, Schmidt NB. Immediate antecedents of marijuana use: an analysis from ecological momentary assessment. J Behav Ther Exp Psychiatry. 2012 Mar;43(1):647-55. doi: 10.1016/j.jbtep.2011.09.010. Epub 2011 Sep 14. PMID 21946296
- [Background] Chen X, Chen P. A comparison of four methods for the analysis of N-of-1 trials. PLoS One. 2014 Feb 4;9(2):e87752. doi: 10.1371/journal.pone.0087752. eCollection 2014. PMID 24503561
- [Background] Centrexion Investigator's Brochure for CNTX-6970. Version 2, 21 February 2019.
- [Background] Ciarleglio A, Petkova E, Ogden T, Tarpey T. Constructing treatment decision rules based on scalar and functional predictors when moderators of treatment effect are unknown. J R Stat Soc Ser C Appl Stat. 2018 Nov;67(5):1331-1356. doi: 10.1111/rssc.12278. Epub 2018 Apr 16. PMID 30546161
- [Background] Dunton GF. Ecological Momentary Assessment in Physical Activity Research. Exerc Sport Sci Rev. 2017 Jan;45(1):48-54. doi: 10.1249/JES.0000000000000092. PMID 27741022
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Edwards RR, Dworkin RH, Turk DC, Angst MS, Dionne R, Freeman R, Hansson P, Haroutounian S, Arendt-Nielsen L, Attal N, Baron R, Brell J, Bujanover S, Burke LB, Carr D, Chappell AS, Cowan P, Etropolski M, Fillingim RB, Gewandter JS, Katz NP, Kopecky EA, Markman JD, Nomikos G, Porter L, Rappaport BA, Rice ASC, Scavone JM, Scholz J, Simon LS, Smith SM, Tobias J, Tockarshewsky T, Veasley C, Versavel M, Wasan AD, Wen W, Yarnitsky D. Patient phenotyping in clinical trials of chronic pain treatments: IMMPACT recommendations. Pain. 2016 Sep;157(9):1851-1871. doi: 10.1097/j.pain.0000000000000602. PMID 27152687
- [Background] Evans K, Romero H, Katz N. Qualitative evaluation and responsiveness of the staircase-evoked pain procedure (STEPP) in two clinical trials of treatments for knee osteoarthritis (OA). https://www.oarsijournal.com/article/S1063-4584(20)30302-2/abstract DOI:https://doi.org/10.1016/j.joca.2020.02.235.
- [Background] Farrar JT, Troxel AB, Haynes K, Gilron I, Kerns RD, Katz NP, Rappaport BA, Rowbotham MC, Tierney AM, Turk DC, Dworkin RH. Effect of variability in the 7-day baseline pain diary on the assay sensitivity of neuropathic pain randomized clinical trials: an ACTTION study. Pain. 2014 Aug;155(8):1622-1631. doi: 10.1016/j.pain.2014.05.009. Epub 2014 May 14. PMID 24831421
- [Background] Gilron I, Ghasemlou N. Chronobiology of chronic pain: focus on diurnal rhythmicity of neuropathic pain. Curr Opin Support Palliat Care. 2014 Dec;8(4):429-36. doi: 10.1097/SPC.0000000000000085. PMID 25111256
- [Background] Gryczynski J, McNeely J, Wu LT, Subramaniam GA, Svikis DS, Cathers LA, Sharma G, King J, Jelstrom E, Nordeck CD, Sharma A, Mitchell SG, O'Grady KE, Schwartz RP. Validation of the TAPS-1: A Four-Item Screening Tool to Identify Unhealthy Substance Use in Primary Care. J Gen Intern Med. 2017 Sep;32(9):990-996. doi: 10.1007/s11606-017-4079-x. Epub 2017 May 26. PMID 28550609
- [Background] Garcia-Palacios A, Herrero R, Belmonte MA, Castilla D, Guixeres J, Molinari G, Banos RM. Ecological momentary assessment for chronic pain in fibromyalgia using a smartphone: a randomized crossover study. Eur J Pain. 2014 Jul;18(6):862-72. doi: 10.1002/j.1532-2149.2013.00425.x. Epub 2013 Nov 22. PMID 24921074
- [Background] Hedeker D, Mermelstein RJ, Demirtas H. An application of a mixed-effects location scale model for analysis of Ecological Momentary Assessment (EMA) data. Biometrics. 2008 Jun;64(2):627-34. doi: 10.1111/j.1541-0420.2007.00924.x. Epub 2007 Oct 26. PMID 17970819
- [Background] Hedeker D, Mermelstein RJ, Demirtas H. Modeling between-subject and within-subject variances in ecological momentary assessment data using mixed-effects location scale models. Stat Med. 2012 Nov 30;31(27):3328-36. doi: 10.1002/sim.5338. Epub 2012 Mar 15. PMID 22419604
- [Background] Hughes CE, Nibbs RJB. A guide to chemokines and their receptors. FEBS J. 2018 Aug;285(16):2944-2971. doi: 10.1111/febs.14466. Epub 2018 Apr 24. PMID 29637711
- [Background] Hunter DJ, Bierma-Zeinstra S. Osteoarthritis. Lancet. 2019 Apr 27;393(10182):1745-1759. doi: 10.1016/S0140-6736(19)30417-9. PMID 31034380
- [Background] Jiang B, Petkova E, Tarpey T, Ogden RT. A Bayesian approach to joint modeling of matrix-valued imaging data and treatment outcome with applications to depression studies. Biometrics. 2020 Mar;76(1):87-97. doi: 10.1111/biom.13151. Epub 2019 Nov 14. PMID 31529701
- [Background] Jung SY, Jang EJ, Nam SW, Kwon HH, Im SG, Kim D, Cho SK, Kim D, Sung YK. Comparative effectiveness of oral pharmacologic interventions for knee osteoarthritis: A network meta-analysis. Mod Rheumatol. 2018 Nov;28(6):1021-1028. doi: 10.1080/14397595.2018.1439694. Epub 2018 Mar 1. PMID 29429391
- [Background] Kalliomaki J, Attal N, Jonzon B, Bach FW, Huizar K, Ratcliffe S, Eriksson B, Janecki M, Danilov A, Bouhassira D; AZD2423 PTN Study Group. A randomized, double-blind, placebo-controlled trial of a chemokine receptor 2 (CCR2) antagonist in posttraumatic neuralgia. Pain. 2013 May;154(5):761-767. doi: 10.1016/j.pain.2013.02.003. Epub 2013 Feb 13. PMID 23523116
- [Background] Kalliomaki J, Jonzon B, Huizar K, O'Malley M, Andersson A, Simpson DM. Evaluation of a novel chemokine receptor 2 (CCR2)-antagonist in painful diabetic polyneuropathy. Scand J Pain. 2013 Apr 1;4(2):77-83. doi: 10.1016/j.sjpain.2012.10.003. PMID 29913894
- [Background] Kan H, Arai Y, Kobayashi M, Nakagawa S, Inoue H, Hino M, Komaki S, Ikoma K, Ueshima K, Fujiwara H, Yokota I, Kubo T. Fixed-flexion view X-ray of the knee superior in detection and follow-up of knee osteoarthritis. Medicine (Baltimore). 2017 Dec;96(49):e9126. doi: 10.1097/MD.0000000000009126. PMID 29245351
- [Background] Koelink PJ, Overbeek SA, Braber S, de Kruijf P, Folkerts G, Smit MJ, Kraneveld AD. Targeting chemokine receptors in chronic inflammatory diseases: an extensive review. Pharmacol Ther. 2012 Jan;133(1):1-18. doi: 10.1016/j.pharmthera.2011.06.008. Epub 2011 Aug 1. PMID 21839114
- [Background] Kroenke K, Krebs EE, Turk D, Von Korff M, Bair MJ, Allen KD, Sandbrink F, Cheville AL, DeBar L, Lorenz KA, Kerns RD. Core Outcome Measures for Chronic Musculoskeletal Pain Research: Recommendations from a Veterans Health Administration Work Group. Pain Med. 2019 Aug 1;20(8):1500-1508. doi: 10.1093/pm/pny279. PMID 30615172
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Li X, Hedeker D. A three-level mixed-effects location scale model with an application to ecological momentary assessment data. Stat Med. 2012 Nov 20;31(26):3192-210. doi: 10.1002/sim.5393. Epub 2012 Aug 3. PMID 22865663
- [Background] Lin WC, Burke L, Schlenk EA, Yeh CH. Use of an Ecological Momentary Assessment Application to Assess the Effects of Auricular Point Acupressure for Chronic Low Back Pain. Comput Inform Nurs. 2019 May;37(5):276-282. doi: 10.1097/CIN.0000000000000478. PMID 31094917
- [Background] Lundeen J, McCall WV, Looney S. Dealing with Methodological Issues in the Functional Data Analysis of Actigraphy Data. Journal of Biometrics & Biostatistics 2019; 10: 429.
- [Background] May M, Junghaenel DU, Ono M, Stone AA, Schneider S. Ecological Momentary Assessment Methodology in Chronic Pain Research: A Systematic Review. J Pain. 2018 Jul;19(7):699-716. doi: 10.1016/j.jpain.2018.01.006. Epub 2018 Jan 31. PMID 29371113
- [Background] McWilliams LA, Kowal J, Wilson KG. Development and evaluation of short forms of the Pain Catastrophizing Scale and the Pain Self-efficacy Questionnaire. Eur J Pain. 2015 Oct;19(9):1342-9. doi: 10.1002/ejp.665. Epub 2015 Mar 11. PMID 25766681
- [Background] MacDonald IJ, Liu SC, Su CM, Wang YH, Tsai CH, Tang CH. Implications of Angiogenesis Involvement in Arthritis. Int J Mol Sci. 2018 Jul 10;19(7):2012. doi: 10.3390/ijms19072012. PMID 29996499
- [Background] Norton S, Cosco T, Doyle F, Done J, Sacker A. The Hospital Anxiety and Depression Scale: a meta confirmatory factor analysis. J Psychosom Res. 2013 Jan;74(1):74-81. doi: 10.1016/j.jpsychores.2012.10.010. Epub 2012 Nov 18. PMID 23272992
- [Background] Osani MC, Vaysbrot EE, Zhou M, McAlindon TE, Bannuru RR. Duration of Symptom Relief and Early Trajectory of Adverse Events for Oral Nonsteroidal Antiinflammatory Drugs in Knee Osteoarthritis: A Systematic Review and Meta-Analysis. Arthritis Care Res (Hoboken). 2020 May;72(5):641-651. doi: 10.1002/acr.23884. Epub 2020 Apr 14. PMID 30908885
- [Background] Park H, Petkova E, Tarpey T, Ogden RT. A single-index model with multiple-links. J Stat Plan Inference. 2020 Mar;205:115-128. doi: 10.1016/j.jspi.2019.05.008. Epub 2019 Jul 4. PMID 32831459
- [Background] Park H, Petkova E, Tarpey T, Ogden RT. A constrained single-index regression for estimating interactions between a treatment and covariates. Biometrics. 2021 Jun;77(2):506-518. doi: 10.1111/biom.13320. Epub 2020 Jul 3. PMID 32573759
- [Background] Parry EL, Thomas MJ, Peat G. Defining acute flares in knee osteoarthritis: a systematic review. BMJ Open. 2018 Jul 19;8(7):e019804. doi: 10.1136/bmjopen-2017-019804. PMID 30030311
- [Background] Perrot S, Lanteri-Minet M. Patients' Global Impression of Change in the management of peripheral neuropathic pain: Clinical relevance and correlations in daily practice. Eur J Pain. 2019 Jul;23(6):1117-1128. doi: 10.1002/ejp.1378. Epub 2019 Mar 18. PMID 30793414
- [Background] Petkova E, Park H, Ciarleglio A, Todd Ogden R, Tarpey T. Optimising treatment decision rules through generated effect modifiers: a precision medicine tutorial. BJPsych Open. 2019 Dec 3;6(1):e2. doi: 10.1192/bjo.2019.85. PMID 31791433
- [Background] Plummer F, Manea L, Trepel D, McMillan D. Screening for anxiety disorders with the GAD-7 and GAD-2: a systematic review and diagnostic metaanalysis. Gen Hosp Psychiatry. 2016 Mar-Apr;39:24-31. doi: 10.1016/j.genhosppsych.2015.11.005. Epub 2015 Nov 18. PMID 26719105
- [Background] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- [Background] Reginster JY, Reiter-Niesert S, Bruyere O, Berenbaum F, Brandi ML, Branco J, Devogelaer JP, Herrero-Beaumont G, Kanis J, Maggi S, Maheu E, Richette P, Rizzoli R, Cooper C. Recommendations for an update of the 2010 European regulatory guideline on clinical investigation of medicinal products used in the treatment of osteoarthritis and reflections about related clinically relevant outcomes: expert consensus statement. Osteoarthritis Cartilage. 2015 Dec;23(12):2086-2093. doi: 10.1016/j.joca.2015.07.001. Epub 2015 Jul 14. PMID 26187570
- [Background] Puljak L, Marin A, Vrdoljak D, Markotic F, Utrobicic A, Tugwell P. Celecoxib for osteoarthritis. Cochrane Database Syst Rev. 2017 May 22;5(5):CD009865. doi: 10.1002/14651858.CD009865.pub2. PMID 28530031
- [Background] Read SJ, Dray A. Osteoarthritic pain: a review of current, theoretical and emerging therapeutics. Expert Opin Investig Drugs. 2008 May;17(5):619-40. doi: 10.1517/13543784.17.5.619. PMID 18447590
- [Background] Salaffi F, Leardini G, Canesi B, Mannoni A, Fioravanti A, Caporali R, Lapadula G, Punzi L; GOnorthrosis and Quality Of Life Assessment (GOQOLA). Reliability and validity of the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index in Italian patients with osteoarthritis of the knee. Osteoarthritis Cartilage. 2003 Aug;11(8):551-60. doi: 10.1016/s1063-4584(03)00089-x. PMID 12880577
- [Background] Salaffi F, Stancati A, Silvestri CA, Ciapetti A, Grassi W. Minimal clinically important changes in chronic musculoskeletal pain intensity measured on a numerical rating scale. Eur J Pain. 2004 Aug;8(4):283-91. doi: 10.1016/j.ejpain.2003.09.004. PMID 15207508
- [Background] Serbina NV, Jia T, Hohl TM, Pamer EG. Monocyte-mediated defense against microbial pathogens. Annu Rev Immunol. 2008;26:421-52. doi: 10.1146/annurev.immunol.26.021607.090326. PMID 18303997
- [Background] Schalet BD, Hays RD, Jensen SE, Beaumont JL, Fries JF, Cella D. Validity of PROMIS physical function measured in diverse clinical samples. J Clin Epidemiol. 2016 May;73:112-8. doi: 10.1016/j.jclinepi.2015.08.039. Epub 2016 Mar 9. PMID 26970039
- [Background] Schmid CH, Duan N. Statistical design and analytic considerations for N-of-1 trials. Design and Implementation of N-of-1 Trials: A User's Guide Rockville, MD: Agency for Healthcare Research and Quality; 2014. p. 33-52.
- [Background] Sullivan MJL, Bishop S, Pivik J. The pain catastrophizing scale: development and validation. Psychol Assess 1995; 7: 432-524.
- [Background] Timmermans EJ, de Koning EJ, van Schoor NM, van der Pas S, Denkinger MD, Dennison EM, Maggi S, Pedersen NL, Otero A, Peter R, Cooper C, Siviero P, Castell MV, Herbolsheimer F, Edwards M, Limongi F, Deeg DJH, Schaap LA. Within-person pain variability and physical activity in older adults with osteoarthritis from six European countries. BMC Musculoskelet Disord. 2019 Jan 5;20(1):12. doi: 10.1186/s12891-018-2392-0. PMID 30611248
- [Background] Treister R, Honigman L, Lawal OD, Lanier RK, Katz NP. A deeper look at pain variability and its relationship with the placebo response: results from a randomized, double-blind, placebo-controlled clinical trial of naproxen in osteoarthritis of the knee. Pain. 2019 Jul;160(7):1522-1528. doi: 10.1097/j.pain.0000000000001538. PMID 30817436
- [Background] Treister R, Suzan E, Lawal OD, Katz NP. Staircase-evoked Pain May be More Sensitive Than Traditional Pain Assessments in Discriminating Analgesic Effects: A Randomized, Placebo-controlled Trial of Naproxen in Patients With Osteoarthritis of the Knee. Clin J Pain. 2019 Jan;35(1):50-55. doi: 10.1097/AJP.0000000000000651. PMID 30222614
- [Background] van Buuren S, Groothuis-Oudshoorn K. Multivariate Imputation by Chained Equations in R. Journal of Statistical Software, 2011, 45(3), 1-67.
- [Background] Wasan AD, Alter BJ, Edwards RR, Argoff CE, Sehgal N, Walk D, Moeller-Bertram T, Wallace MS, Backonja M. Test-Retest and Inter-Examiner Reliability of a Novel Bedside Quantitative Sensory Testing Battery in Postherpetic Neuralgia Patients. J Pain. 2020 Jul-Aug;21(7-8):858-868. doi: 10.1016/j.jpain.2019.11.013. Epub 2019 Dec 11. PMID 31837446
- [Background] White FA, Feldman P, Miller RJ. Chemokine signaling and the management of neuropathic pain. Mol Interv. 2009 Aug;9(4):188-95. doi: 10.1124/mi.9.4.7. PMID 19720751
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Zucker DR, Schmid CH, McIntosh MW, D'Agostino RB, Selker HP, Lau J. Combining single patient (N-of-1) trials to estimate population treatment effects and to evaluate individual patient responses to treatment. J Clin Epidemiol. 1997 Apr;50(4):401-10. doi: 10.1016/s0895-4356(96)00429-5. PMID 9179098
- [Derived] Edwards RR, Tarpey T, Ashburn M, Baer C, Campbell A, Dworkin RH, Gaspard G, Flynn M, Hade E, Jain N, Judge H, Kamp C, Li Y, Meropol S, Petkova E, Philip A, Przkora R, Rathmell JP, Robinson-Papp J, Samuels J, Sehgal N, Sienty J, Stacey B, Wallace M, Wasan AD, Wise B, Yu C, Fava M, Troxel AB. A double-blind, placebo-controlled, multi-crossover trial of treatment with a chemokine antagonist for knee osteoarthritis pain. Pain. 2026 Jan 6. doi: 10.1097/j.pain.0000000000003904. Online ahead of print. PMID 41468282

RESULTS

PARTICIPANT FLOW:
Groups:
- 300mg BID, Then Placebo: Participants initially received 300 mg BID of CNTX-6970 for 6 weeks (Block 1, Period 1). Following this, they were administered matching placebo BID for another 6 weeks (Block 1, Period 2). After a total of 12 weeks, participants received 300 mg BID of CNTX-6970 again for 6 weeks (Block 2, Period 1). Finally, after 18 weeks of total treatment, participants received matching placebo for an additional 6 weeks (Block 2, Period 2), completing a 24-week study period.
- Placebo, Then 300 mg CNTX-6970 BID: Participants initially received placebo BID for 6 weeks (Block 1, Period 1). Following this, they were administered CNTX-6970 BID for another 6 weeks (Block 1, Period 2). After a total of 12 weeks, participants received placebo BID again for 6 weeks (Block 2, Period 1). Finally, after 18 weeks of total treatment, participants received CNTX-6970 BID for an additional 6 weeks (Block 2, Period 2), completing a 24-week study period.
Period: Overall Study
Arm/Group | 300mg BID, Then Placebo | Placebo, Then 300 mg CNTX-6970 BID
Started | 28 | 27 (Multi-crossover study, all participants were randomized to recieve 300 mg CNTX-9670 BID and Placebo)
Completed | 19 | 18 (Multi-crossover study, all participants were randomized to recieve 300 mg CNTX-9670 BID and Placebo)
Not Completed | 9 | 9
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 2 | 4
Not completed — Non compliance | 0 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Stopping criteria met | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Population: Intension-to-Treat (ITT) - All randomized participants
Groups:
- 300mg BID, Then Placebo (DPPD): Participants initially received 300 mg BID of CNTX-6970 for 6 weeks (Block 1, Period 1). Following this, they were administered matching placebo BID for another 6 weeks (Block 1, Period 2). After a total of 12 weeks, participants received 300 mg BID of CNTX-6970 again for 6 weeks (Block 2, Period 1). Finally, after 18 weeks of total treatment, participants received matching placebo for an additional 6 weeks (Block 2, Period 2), completing a 24-week study period.
- Placebo, Then 300 mg CNTX-6970 BID (PDDP): Participants initially received placebo BID for 6 weeks (Block 1, Period 1). Following this, they were administered CNTX-6970 BID for another 6 weeks (Block 1, Period 2). After a total of 12 weeks, participants received placebo BID again for 6 weeks (Block 2, Period 1). Finally, after 18 weeks of total treatment, participants received CNTX-6970 BID for an additional 6 weeks (Block 2, Period 2), completing a 24-week study period.
- Total: Total of all reporting groups
Arm/Group | 300mg BID, Then Placebo (DPPD) | Placebo, Then 300 mg CNTX-6970 BID (PDDP) | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 14 | 33
  >=65 years | 9 | 13 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 19 | 21 | 40
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55
Moderate to severe knee pain stable for 6 months [Count of Participants; unit: Participants] | 28 | 27 | 55
Confirmation of Knee OA by central radiologist [Count of Participants; unit: Participants] | 28 | 27 | 55
Two or more failed therapies [Count of Participants; unit: Participants] | 28 | 27 | 55
mid-high lain score as defined by the WOMAC-A and NRSs [Count of Participants; unit: Participants] | 28 | 27 | 55
BMI less than or equal to 40 [Count of Participants; unit: Participants] | 28 | 27 | 55
Compliant with study requirements before the baseline visit [Count of Participants; unit: Participants] | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC-A)
Description: The primary outcome measure used to assess efficacy will be patient-reported knee pain using the WOMAC Part A (Bellamy, et al., 1988).We will use the numerical rating scale version of the WOMAC, with the subject assessing each of 5 questions using an 11-point (0 to 10) scale; the total score is the sum of the individual item scores (range 0-50). A higher WOMAC score represents worse symptom severity.
Time Frame: 24 Weeks
Population: Intension-to-Treat (ITT) - All randomized participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- 300mg BID CNTX-6970 (DPPD): B1P1: Block 1 Period 1: Participants were instructed to take 300 mg CNTX-6970 BID for weeks 1 through 6
- Placebo BID (DPPD): B1P2: Block 1 Period 2: Participants were instructed to take matching placebo BID for weeks 6 through 12
- Placebo BID (PDDP): B1P1: Block 1 Period 1: Participants were instructed to take matching placebo BID for weeks 1 through 6
- 300 mg BID CNTX-6970 (PDDP): B1P2: Block 1 Period 2: Participants were instructed to take 300 mg CNTX-6970 BID for weeks 6 through 12
- Placebo BID (DPPD): B2P1: Block 2 Period 1: Participants were instructed to take matching placebo BID for weeks 12 through 18
- 300 mg CNTX-6970 (DPPD): B2P2: Block 2 Period 2: Participants were instructed to take 300 mg CNTX-6970 BID for weeks 18 through 24
- 300 mg CNTX-6970 BID (PDDP): B2P1: Block 2 Period 1: Participants were instructed to take 300 mg CNTX-6970 BID for weeks 12 through 18
- Placebo BID (PDDP): B2P2: Block 2 Period 2: Participants were instructed to take matching Placebo BID for weeks 18 through 24
Arm/Group | 300mg BID CNTX-6970 (DPPD): B1P1 | Placebo BID (DPPD): B1P2 | Placebo BID (PDDP): B1P1 | 300 mg BID CNTX-6970 (PDDP): B1P2 | Placebo BID (DPPD): B2P1 | 300 mg CNTX-6970 (DPPD): B2P2 | 300 mg CNTX-6970 BID (PDDP): B2P1 | Placebo BID (PDDP): B2P2
Number analyzed (Participants) | 26 | 21 | 23 | 19 | 20 | 19 | 17 | 16
Score on a scale | 22.5 (12.5) | 18.6 (12.5) | 18.9 (10.1) | 18.2 (11.6) | 18.3 (13.1) | 18.6 (11.9) | 19.4 (9.6) | 16.8 (9.6)
Statistical Analysis 1: Comparison: 300mg BID CNTX-6970 (DPPD): B1P1 vs Placebo BID (DPPD): B1P2 vs Placebo BID (PDDP): B1P1 vs 300 mg BID CNTX-6970 (PDDP): B1P2 vs Placebo BID (DPPD): B2P1 vs 300 mg CNTX-6970 (DPPD): B2P2 vs 300 mg CNTX-6970 BID (PDDP): B2P1 vs Placebo BID (PDDP): B2P2; Null hypothesis is that there was no difference in mean WOMAC-A pain between CNTX-6970 and Placebo. Linear mixed-effect models were used with block, period, sex, age, and KL-grade as covariates and treatment group as factor, with random effects for sites and subjects nested within sites. The test was performed with significance level of 0.05 (two-sided). Power was computed for effect sizes ranging from 0.25 to 0.50 using Monte Carlo simulation, and exceeded 80%; Test type: Superiority; p = .006, Mixed Models Analysis — A 95% confidence interval for the treatment coefficient in the linear mixed-effect model was (-3.033, -0.514), where the reference level was the active treatment; model treatment coefficient = -1.774, 95% CI 2-sided [-3.033 to -0.514], Standard Deviation 0.639

2. Primary Outcome: Treatment Emergent Adverse Events (TEAEs)
Description: The primary safety endpoint is the incidence of treatment emergent adverse events (TEAEs), reported between the administration of study drug on Day 1 and the completion of the study at week 24 or early termination.
Time Frame: 24 Weeks
Population: Intension-to-Treat (ITT) - All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | 300mg BID CNTX-6970 (DPPD): B1P1 | Placebo BID (DPPD): B1P2 | Placebo BID (PDDP): B1P1 | 300 mg BID CNTX-6970 (PDDP): B1P2 | Placebo BID (DPPD): B2P1 | 300 mg CNTX-6970 (DPPD): B2P2 | 300 mg CNTX-6970 BID (PDDP): B2P1 | Placebo BID (PDDP): B2P2
Number analyzed (Participants) | 28 | 25 | 27 | 23 | 20 | 20 | 19 | 17
Participants | 14 | 7 | 14 | 7 | 3 | 4 | 7 | 3

3. Secondary Outcome: Numeric Rating Scale (NRS)
Description: Daily Knee Pain Intensity on a 0-10 Numeric Rating Scale (NRS). Pain intensity is reported by patients with chronic pain as one of the most important targets of treatment, and daily pain intensity ratings are a recommended core outcome measure for clinical trials of treatments for chronic pain. Daily ratings are preferable to ratings of recalled pain over longer time periods such as a week, as daily ratings minimize the influence of recall biases (Dworkin et al., 2005). Participants provide one-daily reports (at the end of the day) of their average knee pain intensity on a 0-10 pain intensity NRS over the course of a week, and those daily ratings are averaged to compute a mean knee pain intensity score. Participants will record their Daily Pain Intensity Numeric Rating Scale (NRS) 0-10 each day for one week prior to each clinic visit using NEForm. Lower NRS values correspond to less pain.
Time Frame: 24 Weeks
Population: Intension-to-Treat (ITT) - All randomized participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 300mg BID CNTX-6970 (DPPD): B1P1 | Placebo BID (DPPD): B1P2 | Placebo BID (PDDP): B1P1 | 300 mg BID CNTX-6970 (PDDP): B1P2 | Placebo BID (DPPD): B2P1 | 300 mg CNTX-6970 (DPPD): B2P2 | 300 mg CNTX-6970 BID (PDDP): B2P1 | Placebo BID (PDDP): B2P2
Number analyzed (Participants) | 21 | 13 | 11 | 15 | 15 | 11 | 11 | 10
units on a scale | 4.8 (2.4) | 3.8 (2.4) | 4.4 (2.3) | 4.3 (2.4) | 3.8 (2.9) | 4.7 (2.2) | 4.5 (2.3) | 3.5 (2.7)

4. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC-C)
Description: WOMAC-C (Function subscale) (Bellamy et al, 1988). The WOMAC-physical function subscale contains 17 items assessing daily functioning, each using an 11-point (0 to 10) numerical rating scale. The total index score (0-170) is the sum of the items. A higher WOMAC function score represents worse functioning and less ability to engage in daily activities.
Time Frame: 24 Weeks
Population: Intension-to-Treat (ITT) - All randomized participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 300mg BID CNTX-6970 (DPPD): B1P1 | Placebo BID (DPPD): B1P2 | Placebo BID (PDDP): B1P1 | 300 mg BID CNTX-6970 (PDDP): B1P2 | Placebo BID (DPPD): B2P1 | 300 mg CNTX-6970 (DPPD): B2P2 | 300 mg CNTX-6970 BID (PDDP): B2P1 | Placebo BID (PDDP): B2P2
Number analyzed (Participants) | 26 | 21 | 23 | 19 | 20 | 19 | 17 | 16
units on a scale | 72.0 (39.9) | 59.8 (41.4) | 58.7 (37.4) | 55.2 (40.2) | 60.4 (44.0) | 63.7 (39.1) | 61.4 (32.9) | 54.9 (36.2)

5. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Anxiety
Description: The HADS is a 14-item self-report questionnaire designed to assess symptoms of anxiety and depression in those with medical illness (Norton et al, 2013). This scale has 14 items, 7 related to anxiety and 7 to depression, rated on 4 points (0 to 3) in domains of intensity or frequency. Scoring is done separately for depression and for anxiety and each domain is interpreted as normal for scores of 0-7, borderline abnormal (borderline case) for scores of 8-10 and abnormal (case) for scores of 11-21. This scale is used to assess depression and anxiety in addition to HEAL/EPPIC-Net core data elements (CDEs) because of its higher sensitivity to change especially in patients with medical illnesses.
Time Frame: 24 Weeks
Population: Participants initially received placebo BID for 6 weeks (Block 1, Period 1). Following this, they were administered CNTX-6970 BID for another 6 weeks (Block 1, Period 2). After a total of 12 weeks, participants received placebo BID again for 6 weeks (Block 2, Period 1). Finally, after 18 weeks of total treatment, participants received CNTX-6970 BID for an additional 6 weeks (Block 2, Period 2), completing a 24-week study period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 300mg BID CNTX-6970 (DPPD): B1P1 | Placebo BID (DPPD): B1P2 | Placebo BID (PDDP): B1P1 | 300 mg BID CNTX-6970 (PDDP): B1P2 | Placebo BID (DPPD): B2P1 | 300 mg CNTX-6970 (DPPD): B2P2 | 300 mg CNTX-6970 BID (PDDP): B2P1 | Placebo BID (PDDP): B2P2
Number analyzed (Participants) | 26 | 21 | 23 | 19 | 20 | 19 | 17 | 16
units on a scale | 2.9 (2.5) | 2.2 (2.4) | 2.8 (2.3) | 1.9 (2.5) | 2.7 (2.6) | 2.2 (2.2) | 1.9 (2.4) | 2.1 (2.4)

6. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The PGIC is a single-item measure of patient-reported improvement that is widely used as a general outcome measure in studies of chronic pain patients, including OA patients (Salaff et al, 2004). It is often used as an index of treatment-associated change, and patient-reported improvements in the form of PGIC scores correlate robustly with significant improvement in pain intensity, pain interference with activities of daily living, mood, and quality of life (Perrot and Lanteri-Minet, 2019).
  The PCIC was collected at baseline and week 24. PGIC is scored from 0-6, where lower values correspond to better outcomes (e.g., 0 = very much improved, whereas 6 is very much worse).
Time Frame: 24 Weeks
Population: Intension-to-Treat (ITT) - All randomized participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo BID (PDDP): B2P2 | 300 mg CNTX-6970 (DPPD): B2P2
Number analyzed (Participants) | 16 | 19
units on a scale | 1.6 (1.2) | 1.8 (1.2)

7. Secondary Outcome: Serum Levels of Cytokines and Chemokines
Description: Assessed at baseline and at the end of each treatment period (weeks 6, 12, 18, and 24).Serum levels are measured in Picograms per millilitre (pg/mL). Analyses were performed for Aim 5 to assess the efficacy of CNTX-6970 (300mg BID) in comparison to placebo in biomarkers from (b) serum and synovial fluid levels of chemokines and cytokines; and (c) Synovial monocyte chemoattractant protein-1/CCR-2 receptor binding inhibition in blood and synovial fluid.
  The following 9 biomarkers had sufficient data based on either the ability to fit models A and/or B and at least 50% of the values were above the minimum detectable threshold:
  Alpha.2.Macroglobulin..A2Macro, Immunoglobulin.A..IgA, Macrophage.Inflammatory.Protein.1.beta..MIP.1.beta, Monocyte.Chemotactic.Protein.1..MCP.1, Serum.Amyloid.P.Component..SAP,
Time Frame: 24 Weeks
Population: Per Protocol: All randomized participants excluding participants with major protocol deviations. Major protocol deviations are those with early terminated from the study and those who had inclusion/exclusion criteria deviation or a treatment dispensing error judged to be significant by study leadership. In this study, only one participant had a treatment dispending error.
Measure: Mean (Standard Deviation); unit: log(pg/mL)
Arm/Group | 300mg BID CNTX-6970 (DPPD): B1P1 | Placebo BID (DPPD): B1P2 | Placebo BID (PDDP): B1P1 | 300 mg BID CNTX-6970 (PDDP): B1P2 | Placebo BID (DPPD): B2P1 | 300 mg CNTX-6970 (DPPD): B2P2 | 300 mg CNTX-6970 BID (PDDP): B2P1 | Placebo BID (PDDP): B2P2
Number analyzed (Participants) | 15 | 16 | 7 | 10 | 15 | 16 | 10 | 11
log(pg/mL)
  Alpha 2 Macroglobulin | 1.0 (0.3) | 1.1 (0.3) | 1.2 (0.2) | 1.2 (0.2) | 1.0 (0.3) | 1.0 (0.3) | 1.2 (0.2) | 1.2 (0.2)
  Immunoglobulin A IgA | 0.4 (1.3) | 0.6 (1.3) | 1.1 (0.4) | 1.0 (0.6) | 0.6 (1.4) | 0.6 (1.5) | 0.9 (0.6) | 0.8 (0.6)
  Serum Amyloid P Component | 2.6 (0.3) | 2.6 (0.2) | 2.6 (0.3) | 2.6 (0.3) | 2.7 (0.2) | 2.6 (0.3) | 2.7 (0.2) | 2.8 (0.3)
  Thyroxine Binding Globulin | 3.8 (0.3) | 3.9 (0.2) | 3.8 (0.2) | 3.9 (0.1) | 3.9 (0.3) | 3.8 (0.3) | 3.9 (0.2) | 3.9 (0.2)
  Vitamin D Binding Protein: number analyzed (Participants) | 15 | 15 | 6 | 9 | 14 | 16 | 9 | 9
  Vitamin D Binding Protein | 5.5 (0.4) | 5.6 (0.3) | 5.5 (0.4) | 5.6 (0.2) | 5.6 (0.4) | 5.6 (0.4) | 5.7 (0.3) | 5.7 (0.4)
  Von Willebrand Factor | 5.1 (0.5) | 5.1 (0.5) | 5.6 (0.2) | 5.1 (0.7) | 5.2 (0.6) | 5.1 (0.6) | 5.3 (0.4) | 5.3 (0.4)
  T Cell Specific Protein RANTES | 2.9 (0.7) | 3.0 (0.5) | 3.0 (0.5) | 3.0 (0.9) | 2.7 (0.9) | 2.9 (0.7) | 3.0 (0.5) | 3.0 (0.7)
  Monocyte Chemotactic Protein 1 | 7.4 (0.6) | 6.1 (0.6) | 6.0 (0.5) | 7.3 (0.7) | 6.0 (0.5) | 7.0 (1.0) | 7.5 (0.7) | 5.9 (0.6)
  Macrophage Inflammatory Protein 1 beta | 7.0 (0.8) | 6.7 (0.8) | 6.4 (0.6) | 6.8 (0.6) | 6.5 (0.7) | 6.9 (0.7) | 6.9 (0.3) | 6.0 (0.8)

8. Secondary Outcome: MCP-1/CCR-2
Description: Monocyte chemoattractant serum protein-1(MCP-1)/CCR-2 receptor binding inhibition by CNTX-6970. This will be assessed at baseline and at the end of each treatment period (weeks 6, 12, 18 and 24).
  The data is measured in pg per mL, the data in analyzed in the natural log of pg per mL, with higher numbers indicating more binding inhibition.
Time Frame: 24 Weeks
Population: ITT - Intention to Treat
Measure: Mean (Standard Deviation); unit: natural log(pg/mL)
Arm/Group | 300mg BID CNTX-6970 (DPPD): B1P1 | Placebo BID (DPPD): B1P2 | Placebo BID (PDDP): B1P1 | 300 mg BID CNTX-6970 (PDDP): B1P2 | Placebo BID (DPPD): B2P1 | 300 mg CNTX-6970 (DPPD): B2P2 | 300 mg CNTX-6970 BID (PDDP): B2P1 | Placebo BID (PDDP): B2P2
Number analyzed (Participants) | 22 | 19 | 22 | 18 | 19 | 17 | 20 | 18
natural log(pg/mL) | 133.8 (246.9) | 0 (0) | 0 (0) | 312.8 (327.7) | 87.4 (380.8) | 140.5 (234.1) | 387.7 (330.7) | 0 (0)

9. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Depression
Description: as for outcome 5
Time Frame: 24 Weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 300mg BID CNTX-6970 (DPPD): B1P1 | Placebo BID (DPPD): B1P2 | Placebo BID (PDDP): B1P1 | 300 mg BID CNTX-6970 (PDDP): B1P2 | Placebo BID (DPPD): B2P1 | 300 mg CNTX-6970 (DPPD): B2P2 | 300 mg CNTX-6970 BID (PDDP): B2P1 | Placebo BID (PDDP): B2P2
Number analyzed (Participants) | 26 | 21 | 23 | 19 | 20 | 19 | 17 | 16
units on a scale | 2.2 (2.1) | 2.0 (2.5) | 1.6 (1.5) | 1.1 (1.2) | 1.6 (2.0) | 2.2 (2.2) | 1.3 (1.4) | 1.4 (1.5)

10. Secondary Outcome: PROMIS - 6A
Description: PROMIS Sleep Disturbance Scale 6A (Yu et al, 2011). Sleep disruption has a bi-directional relationship with chronic pain and is an important secondary outcome to measure in pain trials (Edwards et al, 2016). The Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance short form is a convenient 6-item scale that correlates strongly with the longer forms. It shows greater measurement precision for assessing sleep disturbance than other commonly-used (and much longer) questionnaires such as the Pittsburgh Sleep Quality Index and the Epworth Sleepiness Scale; its brevity and convenience are a major advantage for both research and clinical settings (Yu et al, 2011). 60 is the most commonly used threshold for clinically significant sleep. The PROMIS Sleep Disturbance Scale is expressed as a T-score, with a population mean of 50 and SD of 10. A higher T-score indicates better physical functioning. Possible T scores in this distribution range from 31.7 to 76.1.
Time Frame: 24 Weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | 300mg BID CNTX-6970 (DPPD): B1P1 | Placebo BID (DPPD): B1P2 | Placebo BID (PDDP): B1P1 | 300 mg BID CNTX-6970 (PDDP): B1P2 | Placebo BID (DPPD): B2P1 | 300 mg CNTX-6970 (DPPD): B2P2 | 300 mg CNTX-6970 BID (PDDP): B2P1 | Placebo BID (PDDP): B2P2
Number analyzed (Participants) | 15 | 21 | 13 | 19 | 20 | 19 | 17 | 16
T score | 48.1 (12.0) | 48.8 (10.7) | 45.1 (8.6) | 48.0 (8.4) | 46.9 (8.4) | 48.5 (8.8) | 48.2 (9.0) | 46.4 (8.8)

11. Secondary Outcome: Staircase-evoked Pain Assessment
Description: This procedure consists of stepping fully up and down onto an 8in (20.32cm) high platform with both feet a total of 24 times. The lead leg is alternated between each up/down cycle. Subjects are instructed to use their normal gait for completing this task and are encouraged to complete the task despite increasing pain, without stopping if possible. The procedure is timed, and current knee pain intensity on a 0-10 Numeric Rating Scale (NRS) is assessed immediately before and following the procedure while the subject is in a seated, resting position. Lower values correspond to less pain.
  The NRS from the post-step was analyzed.
Time Frame: 24 Weeks
Population: ITT - Intention to Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 300mg BID CNTX-6970 (DPPD): B1P1 | Placebo BID (DPPD): B1P2 | Placebo BID (PDDP): B1P1 | 300 mg BID CNTX-6970 (PDDP): B1P2 | Placebo BID (DPPD): B2P1 | 300 mg CNTX-6970 (DPPD): B2P2 | 300 mg CNTX-6970 BID (PDDP): B2P1 | Placebo BID (PDDP): B2P2
Number analyzed (Participants) | 25 | 20 | 22 | 18 | 19 | 18 | 16 | 15
units on a scale | 4.9 (2.8) | 3.8 (2.7) | 3.9 (3.0) | 4.4 (2.7) | 3.9 (3.0) | 3.9 (2.6) | 4.8 (2.8) | 4.9 (2.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent through study completion or early withdrawal (24 weeks). If ongoing at the end of the study, the subject was referred for appropriate treatment.
Description: The investigator or designee was required to record all observed and reported AEs at each visit.
  All AEs, serious and not serious, were recorded on the AE eCRF page using appropriate medical terminology. Severity and relationship to study drug were assessed by the investigator as described in the protocol.
  (add in safety populaton)
Groups:
- Placebo BID (DPPD): B2P1: Block 1 Period 1: Participants were instructed to take matching placebo BID for weeks 1 through 6
Arm/Group | 300mg BID CNTX-6970 (DPPD): B1P1 | Placebo BID (PDDP): B1P1 | 300 mg BID CNTX-6970 (PDDP): B1P2 | Placebo BID (DPPD): B1P2 | Placebo BID (DPPD): B2P1 | 300 mg CNTX-6970 (DPPD): B2P2 | 300 mg CNTX-6970 BID (PDDP): B2P1 | Placebo BID (PDDP): B2P2
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/25 | 0/23 | 0/20 | 0/20 | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 1/25 | 1/23 | 0/20 | 0/20 | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 14/28 | 14/27 | 7/25 | 7/23 | 3/20 | 4/20 | 7/19 | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300mg BID CNTX-6970 (DPPD): B1P1 (N=28) | Placebo BID (PDDP): B1P1 (N=27) | 300 mg BID CNTX-6970 (PDDP): B1P2 (N=25) | Placebo BID (DPPD): B1P2 (N=23) | Placebo BID (DPPD): B2P1 (N=20) | 300 mg CNTX-6970 (DPPD): B2P2 (N=20) | 300 mg CNTX-6970 BID (PDDP): B2P1 (N=19) | Placebo BID (PDDP): B2P2 (N=17)
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
chronic myeloid leukaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300mg BID CNTX-6970 (DPPD): B1P1 (N=28) | Placebo BID (PDDP): B1P1 (N=27) | 300 mg BID CNTX-6970 (PDDP): B1P2 (N=25) | Placebo BID (DPPD): B1P2 (N=23) | Placebo BID (DPPD): B2P1 (N=20) | 300 mg CNTX-6970 (DPPD): B2P2 (N=20) | 300 mg CNTX-6970 BID (PDDP): B2P1 (N=19) | Placebo BID (PDDP): B2P2 (N=17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine leukocyte esterase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye laser surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toe operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss diet (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Product after taste (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gate Disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT05025787/Prot_002.pdf
  • Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT05025787/SAP_001.pdf